CLINICAL TRIAL: NCT00855361
Title: A Pharmacokinetic, Pharmacodynamic and Short-term Safety Study of Single and Multiple Day Doses of Rabeprazole Sodium in Neonates and Pre-term Infants With a Corrected Age of Less Than 44 Weeks With a Presumptive Diagnosis of GERD
Brief Title: A Pharmacokinetics, Pharmacodynamics and Safety Study of Rabeprazole in New Born Infants With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014824; RABGRD1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Erosive Gastroesophageal Reflux Disease; Ulcerative Gastroesophageal Reflux Disease; Endoscopy; Pediatrics; GERD; Rabeprazole, Rabeprazole sodium; AcipHex
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

ARMS (1):
- Rabeprazole sodium (Experimental)
  Interventions: Drug: Rabeprazole sodium

INTERVENTIONS:
Drug: Rabeprazole sodium — One single daily dose of rabeprazole sodium 1 mg as a microgranule formulation for up to 28 consecutive days (Part 1), and one single daily dose of rabeprazole sodium 2 or 3 mg as a microgranule formulation for up to 28 consecutive days (Part 2). The study drug will be administered through a nasogastric or orogastric tube.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, pharmacodynamics, and the safety of rabeprazole sodium for the treatment of gastroesophageal reflux disease (GERD) in newborns and pre-term infants.

DETAILED DESCRIPTION:
This is a multi-center Phase I study in newborns and pre-term infants (less than 44 weeks at the time of the first dose). The drug being studied is rabeprazole sodium, the active pharmaceutical ingredient in AcipHex. This study will consist of two parts, Part 1 and Part 2. Each part will consist of three phases, a pre-treatment phase (screening of up to 7 days before the start of treatment), a treatment phase (up to 28 days) and a post treatment phase (at least 14 days, but no more than 21 days after the last dose of study drug). The maximum study length for each patient will therefore be up to 8 weeks. Patients will be monitored patients with a presumptive diagnosis of GERD and who need a feeding tube for enteral alimentation (complete or partial) in place and have been admitted to a newborn intensive care unit or step down unit. The population pharmacokinetics (PK) results together with the pharmacodynamics (ie, pHmetry) data, the safety and tolerability data from Part 1 will be assessed to determine the two dose levels to be studied in Part 2 before the start of dosing. Pharmacokinetics explores how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time. Pharmacodynamics (PD) studies the action or effects a drug has on the body. All patients in Part 1 will require pH monitoring for clinical management and undergo a 24-hour PD assessment (intraesophageal and intragastric pHmetry). At least 12 patients in Part 2 (at least 6 patients from each dose group) will require pH monitoring and undergo the same PD assessment as patients in Part 1. Patients participating in the pHmetry assessment must be in need of this assessment for their clinical management in the opinion of the Principal Investigator. The intraesophageal and intragastric 24-hour pH PD assessment in both Part 1 and Part 2 will be performed at baseline (Day -1) and after the first dose (Day 1) and fifth dose (Day 5). Sampling for single dose blood level PK evaluations will be performed post-dose on Day 1. Sampling blood level evaluations at the presumed steady-state during multiple dosing will be performed on Day 5. Patients' safety will be monitored throughout the study. At the end of the study, or if any patient prematurely discontinues his/her participation in the study, a safety evaluation will be performed at least 14 days, but no more than 21 days, after the final rabeprazole sodium dose. During the course of the study, after consent each patient will have medical history, a physical, length, weight, vital signs, blood chemistry, and urinalysis. Safety from baseline to the End of Study visit (post-treatment phase) will be evaluated by examining incidence, severity and relationship to the study drug and type of Adverse Events (AEs), urinalysis, physical examination and vital signs. Patients will receive rabeprazole sodium as a single daily dose for up to 28 consecutive days. Patients participating in Part 1 will receive 1.0 mg rabeprazole sodium administered by a nasogastric tube. After four patients complete Part 1, their rabeprazole plasma levels will be assessed and the dose may be increased to 2.0 mg rabeprazole sodium. The population PK results, together with the PD (ie, pHmetry) data, safety and tolerability data from Part 1 will be assessed to determine 2 doses in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must need a feeding tube in place for enteral alimentation (complete or partial) and be in a neonatal intensive care unit or step down unit
* Patients participating in the pHmetry assessment must be in need of this assessment
* New born, neonate or pre-term infants less than 44 weeks with a minimum weight of 0.8 kg and with a presumptive diagnosis of GERD
* Patients who have been treated with, or are currently receiving a proton pump inhibitor (PPI), H2-blockers or antacids
* Patients should be generally healthy, other than for the presence of GERD.

Exclusion Criteria:

* A history of or current clinically significant medical illness (excluding GERD, asthma, reactive airway disease or cystic fibrosis-dependant GERD)
* Continuous drip tube feeding with formula or breast milk
* Patients whose mothers are taking PPIs and who are pumping breast milk to be fed to their infants
* Continuous positive airway pressure (CPAP) delivered via nasal prong or oral mask
* Serum concentrations of hepatic transaminases > 3-fold higher than the upper limit of normal for age creatinine values = 106 micromoles/L
* Clinically relevant abnormal laboratory values
* Treatment with full therapeutic doses of sucralfate or any medication that affects gastrointestinal motility such as baclofen, erythromycin, metoclopramide, cisapride, or domperidone
* A history of allergy or sensitivity to PPIs or to their inactive ingredients

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rabeprazole plasma concentrations (Parts 1 and 2) | Up to Day 5
Thioether metabolite plasma concentrations (Parts 1 and 2) | Up to Day 5
The change from baseline in intraesophageal H+ concentration (Parts 1 and 2) | Baseline, Day 5
The change from baseline in intragastric H+ concentration (Parts 1 and 2) | Baseline, Day 5

SECONDARY OUTCOMES:
The number of patients with adverse events as a measure of safety and tolerability | Approximately 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (19):
- United States (10):
  - Orange, California
  - Washington D.C., District of Columbia
  - Augusta, Georgia
  - Maywood, Illinois
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Lansing, Michigan
  - Omaha, Nebraska
  - Brooklyn, New York
  - Toledo, Ohio
- Aachen, Germany
- Poland (4):
  - Bydgoszcz
  - Lublin Poland
  - Odz
  - Poznan
- United Kingdom (4):
  - Barnsley
  - Manchester
  - Preston
  - Sheffield

REFERENCES:
- See also: A Pharmacokinetic, Pharmacodynamic and Short-term Safety Study of Single and Multiple Day Doses of Rabeprazole Sodium in Neonates and Pre-term Infants with a Corrected Age of Less than 44 Weeks with a Presumptive Diagnosis of GERD — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=782&filename=CR014824_CSR.pdf